CLINICAL TRIAL: NCT00625092
Title: Phase I Hyperthermic Intraperitoneal Oxaliplatin for Peritoneal Malignancies
Brief Title: Hyperthermic Intraperitoneal Oxaliplatin for Peritoneal Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS068; 0601M79448 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Peritoneal Cavity Cancer
Keywords: peritoneal cavity cancer
MeSH Terms: interventions — Fluorouracil; Leucovorin; Oxaliplatin; Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hyperthermic Treatment (Experimental): Patients receiving combination of hyperthermic intraperitoneal chemotherapy (HIPC) with oxaliplatin plus intraperitoneal 5-Fu and intraperitoneal leucovorin with peritoneal metastases.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: cytoreductive surgery

INTERVENTIONS:
Drug: fluorouracil — Post-operative day 1 and day 2, 600mg/m^2 intraperitoneal (IP) held for 23 hours
  Other Names: 5-FU
Drug: leucovorin calcium — Day 0 200 mg/m^2 intraperitoneal held for 2 hours
Drug: oxaliplatin — Day 0 hyperthermic intraperitoneal oxaliplatin held for 30 minutes - assigned dose level: Levels 1 through 7 - 300 to 600 mg/m^2
  Other Names: Eloxatin
Procedure: cytoreductive surgery — Day 0 Cytoreductive surgery is a systematic attempt to remove all or nearly all peritoneal nodules.
  Other Names: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hyperthermia therapy kills tumor cells by heating them to several degrees above normal body temperature. Peritoneal infusion of heated and nonheated chemotherapy drugs after surgery may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of hyperthermic intraperitoneal oxaliplatin followed by intraperitoneal leucovorin and fluorouracil in treating patients with peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and optimal dose of hyperthermic intraperitoneal oxaliplatin when administered during cytoreductive surgery and followed by intraperitoneal leucovorin calcium and fluorouracil in patients with peritoneal malignancies.

Secondary

* To determine the outcome of cytoreductive surgery in these patients.
* To determine the time to disease progression and pattern of failure in patients treated with this regimen.
* To determine the 1 and 5 year survival in patients treated with this regimen.
* To compare quality-of-life pre- and post-surgery in these patients.
* To characterize total- and free-platinum pharmacokinetics in the plasma and total platinum in the intraperitoneal space at baseline, during, and after hyperthermic intraperitoneal chemotherapy (HIPC).
* To assess for the presence of genetic polymorphisms in the XDP and XRCC1 DNA repair genes.
* To assess tumor and normal tissue concentrations for total platinum obtained at baseline and immediately after HIPC.

OUTLINE:

* Cytoreductive Surgery: Patients undergo an exploratory laparotomy to remove all tumor nodules from all peritoneal surfaces prior to gastrointestinal anastomoses. An intraperitoneal drain is placed for postoperative intraperitoneal chemotherapy.
* Hyperthermic peritoneal chemotherapy (HIPC): After cytoreductive surgery, but before intestinal anastomosis, patients receive oxaliplatin into the abdomen cavity at approximately 1 liter/min at 41-42º C and held for 30 minutes at the maximum tolerated dose. A heat exchanger maintains the fluid temperature at 44-46º C to maintain the intraperitoneal temperature at 41-42º C. Patients may receive fluid challenges, furosemide, mannitol, or renal dose dopamine to maintain a brisk diuresis at the discretion of the anesthesiologist.
* Intraperitoneal chemotherapy: After HIPC, patients receive leucovorin calcium intraperitoneally through an intraperitoneal drain where it will remain for 2 hours and then drained. Patients then receive fluorouracil intraperitoneally through the intraperitoneal drain on day 1 and remain in the peritoneal fluid for 23 hours and then drained. The infusion will be repeated on day 2.

Blood samples are collected prior to surgery for pharmacogenetic studies and analyzed for the presence of genetic polymorphisms in the XPD and XRCC1 DNA repair genes and the GSTP1 and GSTM1 glutathione-S-transferase enzymes (i.e., XPD, Asp312Asn, XPD K751Q, XRCC1 Arg399GIn, XRCC1 Arg399Q, GSTP1 l105V, and GSTM1 DEL). Blood samples are also collected periodically for pharmacokinetic studies and analyzed for oxaliplatin concentrations. Normal and tumor tissue are collected periodically and analyzed for total platinum concentrations.

Quality of life is assessed at baseline and at 4, 8, and 12 months.

After completion of study treatment, patients are followed every 4 months for 2 years and then every 6 months for at least 5 years.

ELIGIBILITY:
Inclusion criteria:

* Patients must have histologic proof of peritoneal metastases (includes adenomucinosis)
* Complete tumor resection possible (may include liver metastasis if treatable by resection or radiofrequency ablation)
* Patients may have received previous chemotherapy (except peritoneal) and/or immunotherapy. If previous chemotherapy, at least 4 weeks must have passed since last dose.
* Patients may have received previous radiation therapy, however radiation to the large bowel, small bowel and/or stomach will make the patient ineligible for this study.
* Patients must have a Karnofsky performance score of ≥ 80%.
* Adequate hematologic, renal and hepatic function within 14 days of registration defined as:

  * White blood count (WBC) ≥ 3,000
  * platelet count ≥ 70,000,
  * serum bilirubin ≤ 2.0 mg/dL,
  * serum creatinine ≤ 1.5 mg/dL
* Patients must be at least 18 years of age
* Patients must be able to provide informed consent

Exclusion criteria:

* Metastatic disease is present outside the peritoneal cavity
* Diagnosis of mesothelioma
* Grade 2 or higher sensory neuropathy at time of study enrollment
* History of allergic reaction to platinum compounds
* Pregnant or lactating women. Pregnancy is a contraindication for receiving therapy, thus where relevant, patients will be required to use effective birth control. The agents used in this study include those which are pregnancy category D - clear evidence of risk in pregnancy. There is no information on the excretion of agents into breast milk therefore patients must refrain from breastfeeding while receiving study therapy.
* Previous peritoneal chemotherapy.
* Patients with uncontrolled concurrent medical problems (i.e. diabetes mellitus) or history of uncontrolled cardiovascular disease (no history of hospitalization for acute myocardial infarction or congestive heart failure (CHF) within 3 months prior to registration).
* Patients have psychiatric or addictive disorders that preclude obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of hyperthermic intraperitoneal oxaliplatin | 30 Days Post Treatment

SECONDARY OUTCOMES:
Changes in quality-of-life | Baseline and at 4, 8, and 12 months
  Using the Functional Assessment of Cancer Therapy for Colorectal Cancer (FACT-C) and SF-36 (Quality of Life Evaluation in Dialysis Patients) questionnaires, the quality of life following cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPC) will be reported and compared to the preoperative baseline.
Overall survival | 1 Year and 5 Years
Time to Disease Progression | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Tuttle, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States